CLINICAL TRIAL: NCT02596932
Title: Intrapartum Glucose Management Among Women With Gestational Diabetes Mellitus and Its Impact on Neonatal Blood Glucose Levels
Brief Title: Intrapartum Glucose Management Among Women With Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Maureen Hamel, Maureen S. Hamel MD, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 809018
Record Dates: First submitted 2015-10-31; First posted 2015-11-04 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Intrapartum
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tight control (Other): Intervention Standard Care:
  Tight glucose control protocol: Goal maternal blood glucose 70-100, q 1 hour blood glucose checks, insulin treatment started with single maternal blood glucose level > 100mg/dL or < 60 mg/dL
  Interventions: Other: Standard Protocol for intrapartum glucose management
- Less tight control (Experimental): Intervention:
  Less Tight glucose control protocol: Goal maternal blood glucose 70-120, q 4 hour blood glucose checks (unless symptomatic), insulin treatment started with single maternal blood glucose > 120 mg/dL or < 60mg/dL
  Interventions: Other: Experimental Protocol for intrapartum glucose management

INTERVENTIONS:
Other: Standard Protocol for intrapartum glucose management — Tight glucose control protocol: Goal maternal blood glucose 70-100, q 1 hour blood glucose checks, insulin treatment started with single maternal blood glucose level > 100mg/dL or < 60mg/dL
  Other Names: Tight Control
  Arms: Tight control
Other: Experimental Protocol for intrapartum glucose management — Less Tight: Goal maternal blood glucose 70-120, q 4 hour blood glucose checks (unless symptomatic), insulin treatment started with single maternal blood glucose > 120 mg/dL or < 60 mg/dL
  Other Names: Less Tight Control
  Arms: Less tight control

SUMMARY:
Gestational Diabetes Mellitus (GDM) is one of the most common medical complications of pregnancy. Neonatal hypoglycemia is a common and well described complication for infants born to mothers with GDM and diabetes mellitus (DM) and studies have linked intrapartum maternal glucose levels with neonatal hypoglycemia. While guidelines exist to guide practitioners in how to best manage intrapartum maternal glucose levels among Type I and and Type II DM, there is a paucity of data guiding practitioners in the intrapartum management of blood glucose levels for women with GDM, particularly those treated with insulin antepartum. The goal of this project is to compare two protocols of intrapartum glucose management in women with GDM and investigate the impact on neonatal blood glucose levels.

DETAILED DESCRIPTION:
Research objective- To compare "Tight" vs. "Less Tight" intrapartum glucose management

Hypothesis: Neonates born to mothers managed via the "Less Tight" intrapartum glucose management protocol will have lower mean glucose levels in the first 24 hours of life when compared to mean glucose levels among infants born to mothers managed via the "Tight" intrapartum glucose management protocol.

Study Design: Randomized trial

Population: English or Spanish speaking women with a diagnosis of GDM managed at the Diabetes in Pregnancy Program at Women & Infants Hospital, with a plan to deliver at Women & Infants Hospital

Once enrolled, patients will then be randomized to "Tight" or "Less Tight" intrapartum glucose control.

Once admitted to the labor floor for intrapartum management the appropriate power plan for glucose control will be initiated. The specifics of labor management will be left to the discretion of the provider.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking women with a diagnosis of GDM managed at the Diabetes in Pregnancy Program at Women & Infants Hospital, with a plan to deliver at Women & Infants Hospital

Exclusion Criteria:

* Pre-existing DM, multiple gestations, major fetal anomalies anticipated to require NICU admission, planned cesarean delivery, medications known to effect glucose metabolism other than insulin (i.e. metformin)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2016-02; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Mean neonatal blood glucose levels | 24 hours

SECONDARY OUTCOMES:
Neonatal Intensive Care Unit (NICU) admission | Birth of neonate until time of discharge of neonate to home up to 7 days
  Any admission to Neonatal Intensive Care Unit from moment of birth of neonate until time of discharge of neonate to home
Hours in Neonatal Intensive Care Unit (NICU) | Birth of neonate until time of discharge of neonate to home up to 7 days
  Any time spent in Neonatal Intensive Care Unit from moment of birth of neonate until time of discharge of neonate to home
Maternal hypoglycemia | Intrapartum period

CONTACTS AND LOCATIONS:
Overall Officials: Maureen S Hamel, MD, Principal Investigator — Maternal Fetal Medicine
Locations (1):
- Women & Infants Hospital Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hamel MS, Kanno LM, Has P, Beninati MJ, Rouse DJ, Werner EF. Intrapartum Glucose Management in Women With Gestational Diabetes Mellitus: A Randomized Controlled Trial. Obstet Gynecol. 2019 Jun;133(6):1171-1177. doi: 10.1097/AOG.0000000000003257. PMID 31135731